CLINICAL TRIAL: NCT00884169
Title: Study to Investigate the Efficacy and the Safety of M518101 in Psoriasis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maruho Co., Ltd. (Industry)
Responsible Party: R&D Administration Department, Maruho Co.,Ltd ・Kyoto R&D Center
Allocation: Randomized | Masking: Double
Other Study IDs: M518101-EU03
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Last update posted 2010-11-03 (Estimated); Status verified 2010-11

CONDITIONS: Plaque Psoriasis

INTERVENTIONS:
Drug: M518101 — Proper quantity twice a day
Drug: placebo — Proper quantity twice a day

SUMMARY:
This study is to investigate the efficacy and safety of M518101 in male and female plaque psoriasis patients with refractory plaques.

ELIGIBILITY:
Inclusion Criteria:

* Who are able and willing to give signed informed consent
* Who are male or females aged between 18 and 65 years with plaque psoriasis confirmed by the Investigator.
* Who have less than 20% of body surface area (BSA) afflicted with plaques
* Who are neither pregnant nor breast-feeding, nor plan to become pregnant during the study.

Exclusion Criteria:

* Who have a history of allergy to vitamin D3 derivative preparations.
* Who have a history of relevant drug hypersensitivity.
* Who have a history of contact dermatitis induced by a topical medicine.
* Who are pregnant or lactating.
* Who have any renal or hepatic insufficiency, or clinically significant cardiac, renal or hepatic disease.
* Who have clinically relevant history or presence of any disease or surgical history other than psoriasis which is likely to affect the conduct of the study.
* Whose serum calcium levels exceed the upper limit of reference range
* Who have used any investigational medicinal product and/or participated in any clinical study within 24 weeks
* Who have been treated with systemic therapy within 8 weeks
* Who have been treated with biologics within 12 weeks
* Who have been treated with topical therapy during the wash-out and lead-in period.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2009-07; Study Completion 2009-12

PRIMARY OUTCOMES:
Severity of plaque psoriasis

SECONDARY OUTCOMES:
Investigator and Patient overall assessment

CONTACTS AND LOCATIONS:
Locations (1):
- St Thomas' Hospital, London, United Kingdom